CLINICAL TRIAL: NCT00490542
Title: Double-blind, Placebo-controlled Trial of Ziprasidone (Geodon) for the Depressive Mixed State
Brief Title: Safety Study of Ziprasidone (Geodon) for the Depressive Mixed State
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GA128000
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Results first posted 2014-01-08 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Bipolar Disorder; Bipolar Depression; Depression
Keywords: Bipolar Disorder; Major Depression; Clinical pharmacology; Clinical Trial
MeSH Terms: conditions — Bipolar Disorder; Depression; Depressive Disorder, Major | interventions — ziprasidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo arm (Placebo Comparator): Participants were instructed by a physician to take a study drug daily. Dosing instructions began at 40 mg/day and were increased by increments of 20-40 mg weekly weekly based on target symptoms and tolerability with a target range of 80-160 mg/d of ziprasidone. Participants were not informed whether they were receiving sugar pills or Geodon. Participants in this study arm received sugar pills.
  Interventions: Drug: placebo
- Geodon arm (Active Comparator): Participants were instructed by a physician to take a study drug daily. Dosing instructions began at 40 mg/day and were increased by increments of 20-40 mg weekly weekly based on target symptoms and tolerability with a target range of 80-160 mg/d of ziprasidone. Participants were not informed whether they were receiving sugar pills or Geodon. Participants in this study arm received Geodon.
  Interventions: Drug: ziprasidone (Geodon)

INTERVENTIONS:
Drug: ziprasidone (Geodon) — ziprasidone, geodon. Dosing instructions began at 40 mg/day and were increased by increments of 20-40 mg weekly weekly based on target symptoms and tolerability with a target range of 80-160 mg/d of ziprasidone for 6 weeks.
  Arms: Geodon arm
Drug: placebo — Placebo, sugar pill arm. Dosing instructions began at 40 mg/day and were increased by increments of 20-40 mg weekly weekly based on target symptoms and tolerability with a target range of 80-160 mg/d of ziprasidone for 6 weeks.
  Arms: Placebo arm

SUMMARY:
Mixed states in bipolar disorder have long been recognized. Over a century ago, it was argued that mixed states were the most common episodes in manic-depressive illness. A mixed state is defined as a person who is experiencing symptoms of both depression and mania.

Currently, a person must have depression plus 3 or more manic symptoms for the episode to be diagnosed mixed. Using this narrow view, less than 10% of episodes in patients with bipolar disorder would meet criteria for a mixed episode. A broader view requires that the person have at least 2 manic symptoms. Using this broader view, data suggest that about 50% of episodes in bipolar disorder would be diagnosable as mixed states.

Studies suggest that the majority of persons with a depressive mixed state have bipolar disorder type II. Many people who have a mixed state will also have major depression. Even with such high potential rates of mixed episodes in both bipolar disorder and major depression, there have been few studies addressing the issue.

The purpose of this study is to look at how effective Geodon is in treating the depressive mixed state in people with bipolar or major depression. This will be the first clinical trial that is both double-blind and randomized.

DETAILED DESCRIPTION:
We plan on enrolling 25 subjects from each of the four sites. After signing a consent form, subjects will be screened and asked to have a physical and specific safety labs done to make sure they can safely participate in the study. After the screening visit, subjects will be randomly, like a flip of a coin, placed into one of two groups. One group will get the study drug, Geodon. The other group will get placebo, a sugar pill. Neither the doctor nor subject will know in which group the subject has been placed.

Subjects will see the doctor once a week for 6 weeks. During each visit, we will check and treat any side effects. We will ask questions about mood and go through a number of rating scales and assessments that will look at mood and symptoms. Subjects will also fill out questionnaires at each visit to assess their moods and see how the study is going. At the final visit, subjects will have the same physical exam and lab tests done as in the initial visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar disorder type II, or unipolar major depressive disorder
* If female, non-pregnant/non-lactating
* If a sexually active female of reproductive potential, must be using adequate contraception (i.e., oral contraceptives, barrier protection, or prior tubal ligation)
* Currently meets Diagnostic and Statistical Manual, 4th edition (DSM-IV) criteria for a major depressive episode, and presence of 2 or 3 DSM-IV manic criteria, present for the majority of the time during the past week.
* All other baseline psychotropic drugs will be allowed to be continued unchanged. However, if antidepressant use has been initiated in the previous 2 months, or was thought to be contributing to the depressive mixed state, then antidepressant medications would be discontinued 4 weeks before starting the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2006-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nassir Ghaemi, MD, MPH, Principal Investigator — Tufts University
Locations (4):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - Tufts University, Boston, Massachusetts
  - Cambridge Health Alliance, Cambridge, Massachusetts
  - Duke University, Durham, North Carolina

REFERENCES:
- [Derived] Patkar A, Gilmer W, Pae CU, Vohringer PA, Ziffra M, Pirok E, Mulligan M, Filkowski MM, Whitham EA, Holtzman NS, Thommi SB, Logvinenko T, Loebel A, Masand P, Ghaemi SN. A 6 week randomized double-blind placebo-controlled trial of ziprasidone for the acute depressive mixed state. PLoS One. 2012;7(4):e34757. doi: 10.1371/journal.pone.0034757. Epub 2012 Apr 24. PMID 22545088

RESULTS

PARTICIPANT FLOW:
Groups:
- Double-blind Flexible-dose Placebo Arm: Participants in this arm received placebo and were instructed to take it daily for 6 weeks. Participants did not know whether they were taking placebo or ziprasidone (Geodon). Dosing was flexible. Dosing for all subjects was determined based on clinician judgment in an identical manner to dosing in the ziprasidone arm.
- Double-blind Flexible-dose Ziprasidone Arm: Participants in this arm received a flexible dose of ziprasidone and were instructed to take it daily for 6 weeks. Participants did not know whether they were taking placebo or ziprasidone (Geodon). Dosing for all subjects began at 20 mg twice a day and increased to between 80 and 160 mg/day total.
Period: Overall Study
Arm/Group | Double-blind Flexible-dose Placebo Arm | Double-blind Flexible-dose Ziprasidone Arm
Started | 38 | 35
Completed | 31 | 31
Not Completed | 7 | 4
Not completed — Lost to Follow-up | 3 | 0
Not completed — Adverse Event | 3 | 3
Not completed — Lack of Efficacy | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo Arm: Participants in this arm received placebo and were instructed to take it daily for 6 weeks. Participants did not know whether they were taking placebo or ziprasidone (Geodon).
- Geodon Arm: Participants in this arm received Geodon and were instructed to take it daily for 6 weeks. Participants did not know whether they were taking placebo or ziprasidone (Geodon).
- Total: Total of all reporting groups
Arm/Group | Placebo Arm | Geodon Arm | Total
Number analyzed (Participants) | 38 | 35 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 35 | 73
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (12.7) | 39.1 (11.9) | 38.7 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 18 | 17 | 35
Region of Enrollment [Number; unit: participants]
  United States | 38 | 35 | 73

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure Was Change in Montgomery-Asberg Depression Rating Scale (MADRS) Scores Over Weeks Between Groups.
Description: Change in Montgomery-Asberg Depression Rating Scale score was compared between placebo and ziprasidone arms. The MADRS measures severity of depressive symptoms. The MADRS scale is from 0 (min) to 40 (max) with 0 being not depressed at all and 40 being the most severely depressed. 0 is the best outcome and 40 is the worst outcome.
Time Frame: Baseline to 6 weeks
Population: Power analysis, with beta=0.20 and two-tailed alpha=0.05, was based on pilot studies for the mania registration trials which included mixed episodes and assessed MADRS scores. A projected standard error of the mean difference was assumed to be about twice as much as the mean difference (5-15 points), producing a sample size of about 100.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Groups:
- Ziprasidone Arm: Participants in this arm received Geodon and were instructed to take it daily for 6 weeks. Participants did not know whether they were taking placebo or ziprasidone (Geodon).
Arm/Group | Ziprasidone Arm | Placebo Arm
Number analyzed (Participants) | 35 | 38
Scores on a scale | 11.4 [7.101815 to 15.69818] | 5.9 [1.954045 to 9.845955]
Statistical Analysis 1: Comparison: Ziprasidone Arm vs Placebo Arm; Test type: Superiority or Other; Mean Difference (Final Values) = 5.4, 95% CI 2-sided [0.6 to 10.2]

ADVERSE EVENTS:
Arm/Group | Placebo Arm | Geodon Arm
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/35
Other Adverse Events (participants affected / at risk) | 3/38 | 3/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Arm (N=38) | Geodon Arm (N=35)
akathesia (Psychiatric disorders) | 1 (1) | 1 (1)
chest pain (General disorders) | 1 (1) | 0 (0)
sedation (General disorders) | 0 (0) | 2 (2)
migraines (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
One potential limitation in relation to secondary analyses would be sample size. The randomized study design should account for most potential confounding effects, but residual confounding cannot be completely eliminated without larger studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No